CLINICAL TRIAL: NCT04727320
Title: The Clinical Application of Tauroursodeoxycholic Acid in Patients With Liver Fibrosis.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ling Lv
Record Dates: First submitted 2020-12-25; First posted 2021-01-27 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — ursodoxicoltaurine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient+TUDCA (Experimental)
  Interventions: Drug: Tauroursodeoxycholic acid
- patient+placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tauroursodeoxycholic acid — Oral TUDCA, once a day, one tablet (250mg) at a time for 6 months
  Arms: patient+TUDCA
Drug: Placebo — Oral placebo, once a day, one tablet at a time for 6 months
  Arms: patient+placebo

SUMMARY:
This study is a prospective study. We signed an informed consent form with patients with liver fibrosis and took tauroursodeoxycholic acid orally for half a year. After half a year, liver biopsy was performed using histopathology, immunohistochemistry, and polymerase chain reaction, Western blotting method was used to determine the expression level of fibrosis-related markers to verify the effect of taurodeoxycholic acid on patients with liver fibrosis.

DETAILED DESCRIPTION:
Tauroursodeoxycholic acid is an effective component of bear bile, which has obvious curative effects in the treatment of gallstones and liver diseases. In recent years, the research field of tauroursodeoxycholic acid has been very active, and its chemical synthesis has also attracted much attention. The usage is swallowing with water before going to bed at night. It must be taken regularly, one capsule at a time (250mg), once a day. After 6 months of continuous use, liver biopsy was performed after 6 months. Telling the patient to swallow with water before going to bed at night. It must be taken regularly, one capsule at a time (250mg), once a day. After 6 months of continuous use, liver B-ultrasound biopsy was performed to observe the effect.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of liver cirrhosis and liver fibrosis in patients requiring medical treatment.

Exclusion Criteria:

* Patients with end-stage cirrhosis, liver failure, etc. who need liver transplantation.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-05 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Liver biopsy | up to 24 weeks
  Synthesis of liver extracellular matrix（Synthesis, degradation）

SECONDARY OUTCOMES:
Liver ultrasound | up to 24 weeks
  Liver parenchymal echo（Normal, dense, thickened）